CLINICAL TRIAL: NCT04806867
Title: Selection of Patients With Chronic Inflammatory Rheumatism Requiring Management During the COVID-19 Pandemia Through an Innovative Organizational Strategy
Brief Title: Selection of Patients With Chronic Inflammatory Rheumatism Requiring Management During the COVID-19 Pandemia
Acronym: SePaRIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20_0044 (SePaRIC)
Record Dates: First submitted 2020-12-09; First posted 2021-03-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Inflammatory Rheumatism; Rheumatoid Arthritis; Spondyloarthritis; Inflammatory Arthritis
Keywords: Chronic Inflammatory Rheumatism - COVID-19
MeSH Terms: conditions — COVID-19; Rheumatic Fever; Arthritis, Rheumatoid; Spondylarthritis; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SePaRIC-Covid19 cohort — All patients with Chronic Inflammatory Rheumatism who were contacted by telephone as part of the innovative organizational strategy and who did not object to the use of their data.

SUMMARY:
The project proposes to evaluate a strategy for prioritizing teleconsultation for patients with chronic inflammatory rheumatic diseases during the COVID-19 pandemia. This selection will be done through telephone contact by medical students, supervised by residents and rheumatologists on a patient database. The other objectives are to assess the impact of the pandemia on the physical and mental health of patients classified as being at risk

DETAILED DESCRIPTION:
The COVID-19 pandemic led to the suspension of consultations and hospitalization of the majority of patients followed in the Rheumatology Department of the Limoges University Hospital.

The department therefore implemented a strategy for the management of patients with chronic inflammatory rheumatism (CIR) during this period, which allowed maintaining contact with patients in the patient database.

During this telephone call, an CIR-Covid19 questionnaire was fulfilled in order to prioritize patients requiring rapid management.

The strategy is based on the use of the available health reserve, i.e. volunteered medical students to provide patient management assistance. These students were trained with face-to-face learning in the rheumatology department given by residents on chronic inflammatory rheumatism to remind them of all the elements of diagnosis and management. They had an interview with a senior rheumatologist from the Department to present the questionnaire and its objectives , to give them advice regarding communication with patients, as well as information about the COVID-19 infection and recommendations of the French Rheumatology Society for CIR patients. The students were trained with quizzes on practical situations, with feedback on the answers.

The information's collected in the questionnaire were based on the patients' feelings. Telephone communication does not allow an assessment of disease activity according to validated criteria as it requires a clinical examination.

The opinion of the referring rheumatologist was requested by the patients or by the medical student at the end of the telephone call, depending on the information collected. At any time, the medical students could call upon to senior doctors from the department or residents in case of difficulties.

943 patients were thus contacted between 14/04/2020 and 28/04/2020. They were able to benefit from an optimized management according to the context of the COVID19 pandemic.

These questionnaires were analyze in order to assess the need for specialized follow-up during this period and to evaluate the impact of COVID19 on this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic inflammatory rheumatism who answered the RIC-COVID19 survey during the telephone call set up by the Rheumatology Department of the Limoges University Hospital during the confinement.

Exclusion Criteria:

* Patients objecting to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic inflammatory rheumatism
Sampling Method: Non-Probability Sample
Enrollment: 918 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring an advice from the referring rheumatologist following the telephone survey. | 2 months
  Number of request for advice from the referring Rheumatologist by the student and/or the patient

SECONDARY OUTCOMES:
Evaluate the association between rheumatologist advice asked by student and/or patient and the factors studied | 2 months
  Request for an advice from the referring rheumatologist by the student and/or the patient and the factors studied.
  Factors studied:
  Sex, age, department of residence, RA or AS COVID-19 symptoms, increase in CIR activity, increase in pain, discontinuation of treatment, increase in stress and anxiety, increase in depression, increase in fatigue, increase in sleep disorders, fear of coming to consultation or hospitalization, adaptability with their rheumatic disease, medical loneliness.
COVID-19 infection evaluation in the monitored patient population | 2 months
  Evaluate the proportion of COVID-19 infection in patients monitored in the Rheumatology department at Limoges University Hospital Proportion of COVID-19 serological tests performed and their positivity in this patient population.
Proportion of patients informed about COVID-19 | 2 months
  Evaluate the proportion of patients having received medical information about the Covid-19 pandemic.
Evaluate the association between the increase in rheumatic activity perceived by patients and the factors studied | 2 months
  Evaluate the association between the increase in rheumatic activity perceived by patients and the factors studied using numerical scale of satisfaction following this call from patients and students (0-10) 0: unsatisfied, 10 : fully satisfied
Evaluate the association between pain increase perceived by patients and the factors studied | 2 months
  Percentage increase in pain perceived by patients during the epidemic and factors studied, evaluated by numerical scale during the phone call 0% to 100% (0% represente no pain, and 100% maximal pain)
Evaluate the association between rheumatologist advice asked by student and the factors studied | 2 months
  request for an advice from the referring rheumatologist by the student and the factors studied
Evaluate the association between rheumatologist advice asked by patient and the factors studied | 2 months
  request for an advice from the referring rheumatologist by the patient and the factors studied.
To evaluate the satisfaction of the telephone call with patients and students. Time Frame: phone call day | 2 months
  Numerical scale of satisfaction following this call from patients and students (0-10) 0: unsatisfied, 10 : fully satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Pascale PV Vergne-Salle, MD-PhD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Service de Rhumatologie, CHu de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: Undecided